CLINICAL TRIAL: NCT01342393
Title: Proof of Concept Study for First-Sight Refractive Error Correction:Direct Comparison to Manifest Refraction and Autorefraction Results
Brief Title: Proof of Concept Study for First-Sight Refractive Error Correction: Direct Comparison to Manifest Refraction and Autorefraction Results
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 131-11
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Proof of concept study is to compare the best corrected visual acuity obtained via First-Sight lenses with the clinical "gold standard" of manifest refraction and autorefraction.

DETAILED DESCRIPTION:
Uncorrected refractive error is a frequent cause of visual impairment in the global population. In 2006, the World Health Organization released global estimates on visual impairment. According to their findings, there are approximately 314 million people in the world whose vision is impaired. Of this population 90% of those individuals live in developing countries and 153 million cases are believed to be due to uncorrected refractive error. The impact of uncorrected refractive error is great, including, but not limited to, loss of employment opportunities, inability to care for family, and inability to receive an education. The challenge is to determine the most effective and accessible method of detecting refractive error and dispensing spectacles for better vision.

In the clinical setting, refractive error is corrected by prescribing spectacles or contact lenses on a daily basis. Typically the patient will first undergo autorefraction, in which a computer-controlled machine is used to objectively calculate the refractive error present as a starting point for the subjective refraction test. This machine, however, is cumbersome and not easily transportable abroad. Typically the machine is held up to the patient's forehead and they are asked to look into the machine at a distant object. While they are looking at this object the machine calculates the refractive error. Next, the patient undergoes manifest refraction, a subjective refractive test that requires the use of trial lenses and patient responses to improve the results calculated by autorefraction, resulting in the best corrected visual acuity for that patient and a prescription for the patient to receive spectacles tailored to their need.

As a testimony to how prevalent uncorrected refractive error is in the developing world, refractive error in Nigerian adults and the prevalence of spectacle use was studied. In an article titled Refractive errors in Nigerian adults: prevalence, types and spectacle coverage, researchers looked at types of refractive errors and the ability of off the shelf spectacles to meet the corrective need in the 13,599 Nigerian adults. Patients underwent autorefraction and a detailed clinical exam and it was discovered that uncorrected refractive errors were responsible for 77.9% of visual impairment at the 20/40 to 20/60 level, and 57.1% at the 20/60 to 20/200 level. It also found that spectacles could improve the vision of 1,279 adults in the 20/40 range and 882 participants at the 20/60 level. However, only 3-4% of those individuals wore spectacles.

First-Sight is a simplified way to correct refractive error. It is easily portable, making it accessible to remote areas of the world. Unlike the study cited above, First-Sight can be brought to remote areas where clinics are not available and patients are not able to afford to pay for the clinic visit. As it is a simplified technique, local health care workers may easily be able to learn how to use First-Sight and dispense spectacles to those in need. Lastly, the sponsor of First-Sight will provide the refracting kits and custom-made spectacles at no cost to the health care workers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 19 years of age and older.
* A refractive error of -4.50 to +4.50 diopter spherical error and astigmatism up to -1.50 diopters on manifest refraction and autorefraction as documented in the patient's medical records.
* Best corrected visual acuity (BCVA) of 20/20 with manifest refraction.
* No known ocular pathology from previous clinical exams that may limit best corrected visual acuity.

Exclusion Criteria:

* Refractive error greater than -4.50 or +4.50 diopter, or astigmatism greater than -1.50 diopters.
* Known ocular (corneal, lenticular, vitreal, or retinal) pathology that may limit BCVA.
* Best corrected visual acuity with spectacles of 20/25 or worse.
* Any previous surgical or laser procedures that may limit BCVA
* 18 years of age and younger

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population with refractive error between -4.50 to +4.50 diopter spherical error and astigmatism up to -1.50 diopters
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Feilmeier, MD, Principal Investigator — UNMC Department of Ophthalmology and Visual Sciences
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmology, Omaha, Nebraska, United States